CLINICAL TRIAL: NCT02957448
Title: An Open-Label, Single-Sequence Study to Evaluate the Effect of Rifampin on the Single-dose Pharmacokinetics of BMS-986141 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Rifampin on the Single-dose Pharmacokinetics (PK) of BMS-986141 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CV006-029
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Atherothrombotic Diseases
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS 986141 and Rifampin (Experimental)
  Interventions: Drug: BMS 986141; Drug: Rifampin

INTERVENTIONS:
Drug: BMS 986141 — Two single doses BMS 986141 (days 1 and 13) and single daily doses Rifampin (days 7-22)
Drug: Rifampin — Two single doses BMS 986141 (days 1 and 13) and single daily doses Rifampin (days 7-22)

SUMMARY:
This study is to evaluate the effect of multiple doses of rifampin on the single-dose PK of BMS 986141 with parameters like Cmax, AUC(INF), AUC(0-T), AUC(0-144h)

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Healthy men and women (not of child bearing potential) as determined by medical history, surgical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests including coagulation parameters.
3. Subjects with body mass index of 18 to 32 kg/m2, inclusive.
4. Women participants must have documented proof that they are not of childbearing potential.
5. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment plus 5 half-lives of Rifampin (1 day) plus 90 days for a total of 91 days post-treatment completion.

Exclusion Criteria:

1. Acute or chronic medical illness, subjects with bleeding diathesis, gastroesophageal reflux disease, gastrointestinal ulcer, hepatic disease,coagulation disorder,dyspepsia and being reliant on contact lenses for vision for the duration of study treatment and for 2 days after discontinuation of study treatment (eyeglasses are allowed).
2. History of nausea, diarrhoea, recent surgery, use of tobacco or nicotine containing products, drug or alcohol use, periodontal disease, hemorrhoids with rectal bleeding and recent blood donation.
3. Prior exposure to BMS-986141 or prothrombin complex, any investigational product or placebo within 4 weeks of study treatment start, any prescription or over the counter drugs except those cleared by BMS clinical monitor.
4. History of hypersensitivity to BMS 986141, rifampin, any rifamycins or related compounds, or any component of the formulations
5. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECGs, or clinical laboratory determinations beyond what is consistent with the target population

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986141 | Days 1-22
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-986141 | Days 1-22
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of BMS-986141 | Days 1-22
Area under the plasma concentration-time curve from time zero to 144 hours postdose (AUC(0-144h)) of BMS-986141 | Days 1-22

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and death | Screening- until 30 days after discontinuation of dosing or subject's participation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx